CLINICAL TRIAL: NCT06634407
Title: Transcatheter Closure of Patent Ductus Arteriosus. Experience of Pediatric Cardiology Unit-Assiut University Hospital
Brief Title: Outcome of Transcatheter Closure of Patent Ductus Arteriosus in Pediatric Cardiology Unit in 3 Years Duration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bassem Eldaba Hosny Fares, pediatric resident, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Transcatheter closure of PDA
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Patent Ductus Arteriosus (PDA)
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDA patients (Other)
  Interventions: Procedure: transcatheter closure

INTERVENTIONS:
Procedure: transcatheter closure — using transcatheter closure of PDA to detect outcome of patients with PDA

SUMMARY:
Transcatheter Closure of Patent Ductus Arteriosus to evaluate the outcome of percutaneous transcatheter closure of patent ductus arteriosus in children

ELIGIBILITY:
Inclusion Criteria:

* Children with Patent Ductus Arteriosus confirmed by echocardiography
* aged from 6 months to 16 years underwent percutaneous transcatheter PDA closure at Pediatric Cardiology Unit.

Exclusion Criteria:

* Children with PDA younger than 6 months or older than 16 years and that are not candidate for transcatheter closure .

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-10-25 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
outcome of trancathter PDA closure | 3 years
  outcome of 90 patients with trancatheter PDA closure in pediatrics using post procedure catheter and echocardiography